CLINICAL TRIAL: NCT01671358
Title: Comparison of Contamination Rates of Medication Storage Cabinets Between Isolation and Non-isolation Rooms With Methicillin-resistant Staphylococcus Aureus (MRSA)
Brief Title: Comparison of Bacterial Contamination Rates Between Isolation and Non-isolation Rooms
Status: Completed | Type: Observational
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Michael Sweet, Pharmacy Clinical Specialist - Quality Outcomes, West Virginia University
Other Study IDs: WVU-00010
Record Dates: First submitted 2012-08-16; First posted 2012-08-23 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus
Keywords: MRSA; Contamination; Isolation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Isolation Rooms for MRSA: Rooms that currently have a patient in them that are in isolation status due to MRSA
- Non-isolation rooms: Rooms that have not been occupied by a patient in isolation due to MRSA for 14 days

SUMMARY:
This study is to determine if medication cabinets located outside of isolation rooms in hospitals and their contents, particularly medications and the delivery folders are at a higher risk of having harmful bacteria on them.

DETAILED DESCRIPTION:
Studies show high touch areas maybe contaminated with organisms such as Methicillin-resistant Staphylococcus aureus(MRSA) and vancomycin-resistant enterococci. MRSA can live on hospital surfaces for 9-14 days. Patients in rooms that were previously MRSA isolation rooms are at higher risk for developing a hospital-acquired infection.

This study is to determine if medication cabinets located outside of MRSA isolation rooms and their contents, particularly medications and the pharmacy delivery folders are at a higher risk of having MRSA colonization on them. This study will use conventional methods to determine if MRSA colonization is present and compare results between non-isolation and isolation rooms. This will evaluate if alternate measures for the reduction of MRSA colonization are needed for the MRSA isolation rooms in regards to medication delivery and storage.

ELIGIBILITY:
Inclusion Criteria:

* Patient rooms with isolation status for MRSA
* Patient rooms without isolation status for MRSA for 14 days

Exclusion Criteria:

* Rooms without medication cabinets directly outside the room

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inaptients at an academic medical center
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Presence of MRSA colonization | Hospital stay, an expected average of 14 days
  Swabbing of four areas of the medication cabinet will be performed (keypad, handle, medication folder and a medication). A Semi-quantitative sampling technique will be used to collect the samples. A sterile saline moistened sterile cotton tip swab will be used to swab the specified areas. The swabs will then be used to inoculate sheep blood agar plates in 4 quadrants. The plates will be incubated for 48 hours. The number of quadrants with growth will be identified. Individual colonies will be removed from the plate with an inoculation loop, then streaked onto a second sheep blood agar plate. The second plates will be incubated for 48 hours. The colonies will then be run through standard identification tests to determine if the colonies are MRSA or not. A comparison will be made between non-isolation and isolation rooms.

SECONDARY OUTCOMES:
Quantification of MRSA colonization | Hospital stay, an expected average of 14 days
  Swabbing of four areas of the medication cabinet will be performed (keypad, handle, medication folder and a medication). A Semi-quantitative sampling technique will be used to collect the samples. A sterile saline moistened sterile cotton tip swab will be used to swab the specified areas. The swabs will then be used to inoculate sheep blood agar plates in 4 quadrants. The plates will be incubated for 48 hours. The number of quadrants with growth will be identified. A comparison between the sites of swabbing will be performed.

OTHER OUTCOMES:
Presence of other bacterial colonization | Hospital stay, an expected average of 14 days
  Swabbing of four areas of the medication cabinet will be performed (keypad, handle, medication folder and a medication). A Semi-quantitative sampling technique will be used to collect the samples. A sterile saline moistened sterile cotton tip swab will be used to swab the specified areas. The swabs will then be used to inoculate sheep blood agar plates in 4 quadrants. The plates will be incubated for 48 hours. The number of quadrants with growth will be identified. Individual colonies will be removed from the plate with an inoculation loop, then streaked onto a second sheep blood agar plate. The second plates will be incubated for 48 hours. The colonies will be categorized as gram negative, gram positive catalase negative, Gram positive coagulase negative Staphylococcus species or methicillin-sensitive Staphylococcus aureus. This will serve as a baseline epidemiology of the hospital and generate other possible hypotheses.
Correlation between MRSA and active infection or colonization of patient | Hospital stay, an expected average of 14 days
  The patient from the same time frame in the rooms sampled and positive for MRSA colonization will be reviewed to determine if they had active infection or were previously colonized.
Correlation between colonization of other positive organisms and active infection or colonization of patient | Hospital stay, an expected average of 14 days
  The patient from the same time frame in the rooms sampled and positive for non-MRSA colonization will be reviewed to determine if they had active infection or were previously colonized.

CONTACTS AND LOCATIONS:
Locations (1):
- West Virginia University Hospitals, Morgantown, West Virginia, United States

REFERENCES:
- [Background] Bures S, Fishbain JT, Uyehara CF, Parker JM, Berg BW. Computer keyboards and faucet handles as reservoirs of nosocomial pathogens in the intensive care unit. Am J Infect Control. 2000 Dec;28(6):465-71. doi: 10.1067/mic.2000.107267. PMID 11114617
- [Background] Sexton T, Clarke P, O'Neill E, Dillane T, Humphreys H. Environmental reservoirs of methicillin-resistant Staphylococcus aureus in isolation rooms: correlation with patient isolates and implications for hospital hygiene. J Hosp Infect. 2006 Feb;62(2):187-94. doi: 10.1016/j.jhin.2005.07.017. Epub 2005 Nov 14. PMID 16290319
- [Background] Oie S, Hosokawa I, Kamiya A. Contamination of room door handles by methicillin-sensitive/methicillin-resistant Staphylococcus aureus. J Hosp Infect. 2002 Jun;51(2):140-3. doi: 10.1053/jhin.2002.1221. PMID 12090803
- [Background] Huang SS, Datta R, Platt R. Risk of acquiring antibiotic-resistant bacteria from prior room occupants. Arch Intern Med. 2006 Oct 9;166(18):1945-51. doi: 10.1001/archinte.166.18.1945. PMID 17030826
- [Background] Huang R, Mehta S, Weed D, Price CS. Methicillin-resistant Staphylococcus aureus survival on hospital fomites. Infect Control Hosp Epidemiol. 2006 Nov;27(11):1267-9. doi: 10.1086/507965. Epub 2006 Sep 28. PMID 17080391